CLINICAL TRIAL: NCT02289547
Title: Randomized Phase 3 Study of Xelox(Capecitabine Plus Oxaliplatin) Followed by Maintenance Capecitabine or Observation in Patients With Advanced Gastric Adenocarcinoma
Brief Title: Phase 3 Study of Xelox Followed by Maintenance Capecitabine in the Advanced Gastric Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Byoungyong Shim, Associated professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMCGA1 Trial
Record Dates: First submitted 2014-10-30; First posted 2014-11-13 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Stomach Neoplasms
Keywords: chemotherapy; stomach neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (No Intervention): observational arm
- Group B (Experimental): arm of capecitabine maintenance treatment
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — maintenance capecitabine therapy after six cycles of XELOX
  Other Names: Xeloda
  Arms: Group B

SUMMARY:
XELOX regimen had a more favorable toxicity profile compared to cisplatin for patients with advanced gastric cancer. The safety profile of oxaliplatin makes it an ideal candidate for combination therapy. However, oxaliplatin induce sensory neuropathy, a cumulative, dose-related toxicity. It may therefore be possible to devise capecitabine maintenance regimen which achieves maximum treatment effect before cumulative neurotoxicity appears. We study that randomized Phase III study of Xelox (Capecitabine plus Oxaliplatin) followed by maintenance Capecitabine or Observation in the gastric cancer patients of stable disease after 6 cycle 1st line of XELOX chemotherapy .

DETAILED DESCRIPTION:
Study rationale : Park et al. observed the oxaliplatin as part of XELOX regimen had a more favorable toxicity profile compared to cisplatin for patients with advanced gastric cancer. The safety profile of oxaliplatin makes it an ideal candidate for combination therapy. However, oxaliplatin induce sensory neuropathy, a cumulative, dose-related toxicity. The response with XELOX regimen generally occurs earlier. It may therefore be possible to devise capecitabine maintenance regimen which achieves maximum treatment effect before cumulative neurotoxicity appears. This regimen was studied in colon and breast cancer.

- Objective: Primary: To evaluate progression free survival Secondary: To evaluated overall survival, response rate, toxicity profile of chemotherapy, quality of life

* Design :Multicenter randomized controlled phase III open label trial Study subjects will be randomized to two groups in a ratio of 1:1 Subjects More than stable disease after 6 cycle 1st line of XELOX chemotherapy (OR non-complete response/non-progressive disease in cases of non-measurable disease before XELOX chemotherapy),
* Treatment Groups Group A : Capecitabine: Capecitabine 1000mg/m2 bid D1-14, q 3 week Group B : Observation
* Evaluation of response and toxicity A response will be evaluated radiologically every two cycles thereafter, or when progression is suspicious by RECIST criteria version 1.1.

A progression-free survival is defined as the time from the date of randomization to the date of first documented disease progression or death due to any cause.

An overall survival is defined as the time from the 1stdate of chemotherapy to the date of death.

Safety will be evaluated every treatment by NCI-CTCAE version 4.0.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven gastric cancer
* Minimum age of 18 years
* Stage IV (regardless of the presence or absence of measurable disease by RECIST criteria) or recurrent after curative surgery
* Negative expression (0, 1) of Her2 Immuno-histochemistry or negative amplification of FISH in Her2 Immuno-histochemistry 2+
* More than stable disease after 6 cycle 1st line of XELOX chemotherapy (OR non-Complete response/non-Progressive disease in cases of non-measurable disease before XELOX chemotherapy)
* Eastern Cooperative Oncology Group Performance status 0-2
* Adequate bone marrow function: Absolute neutrophil count ≥ 1,500/ul, Hemoglobin ≥ 8 g/dL, platelet ≥ 100,000/μl
* Adequate renal function: Serum creatinine ≤ 1.5 x ULN (upper normal limit) or creatinine clearance ≥ 60 ml/min
* Adequate hepatic function: serum bilirubin ≤ 2.5 x UNL, AST and ALT ≤ 2.5 x UNL (≤ 5 x ULN in the presence of liver metastasis)
* Patients must sign an informed consent indicating that they are aware of the investigational nature of the study in keeping with the policy of the hospital

Exclusion Criteria:

* Patients who were exposed previously to any chemotherapy except XELOX for advanced disease
* Patients who received R0 or R1 resection for metastatic or recurrent gastric cancer and without evaluable/measurable disease
* Disease relapsed during or within 4 months after adjuvant therapy
* Patients who had central nervous system and meningeal metastases
* Patients with significant neurologic or psychiatric disorders
* Patients with active infection, severe heart disease, uncontrollable hypertension or diabetes mellitus, myocardial infarction during the preceding 6 months, pregnancy, or breast feeding
* Any previous or concurrent malignancy except for adequately treated non-melanoma skin cancer, in situ cancer of uterine cervix, non-muscle invasive bladder cancer or malignancy without evidence of recurrence within 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From date of randomization until the date of first documented progression, whichever came first, assessed up to 2 years
  every two cycles (6 weeks) until 18 weeks and then every 4 cycles (12 weeks) until progression

SECONDARY OUTCOMES:
Overall survival | From date of randomization until the date of death from any cause, whichever came first, assessed up to 2 years
  every two cycles (6 weeks) until 18 weeks and then every 4 cycles (12 weeks) until death
quality of life in patients measured by QLQ-c30 and STO-22 | From date of randomization until the date of first documented progression, whichever came first, assessed up to 2 years
  every two cycles (6 weeks) until 18 weeks and then every 4 cycles (12 weeks) until progression
Toxicity profile of each patients measured by NCI-CTCAE ver 4.0 | From date of randomization until the date of first documented progression, whichever came first, assessed up to 2 years
  every two cycles (6 weeks) until 18 weeks and then every 4 cycles (12 weeks) until progression

CONTACTS AND LOCATIONS:
Overall Officials: Byoungyong Shim, M.D.,Ph.D, Principal Investigator — St.Vincent's Hospital of The Catholic University of Korea; Young Seon Hong, M.D.,Ph.D, Principal Investigator — Seoul St. Mary's Hopital of The Catholic Univerisity of Korea; In Sook Woo, M.D.,Ph.D, Principal Investigator — St. Mary's Hospital of The Catholic University of Korea; Jae Ho Byun, M.D.,Ph.D, Principal Investigator — Incheon St. Mary's Hopital of The Catholic Univerisity of Korea; Cuk Jin Lee, M.D.,Ph.D, Principal Investigator — Bucheon St. Mary's Hopital of The Catholic Univerisity of Korea; Ji Chan Park, M.D.,Ph.D, Principal Investigator — Daejeon St. Mary's Hopital of The Catholic Univerisity of Korea; Yoon Ho Ko, M.D.,Ph.D, Principal Investigator — Ujeongbu St. Mary's Hopital of The Catholic Univerisity of Korea; Keun Wook Lee, M.D.,Ph.D, Principal Investigator — Bundang Seoul National Hospital
Locations (8):
- South Korea (8):
  - St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Buchon St. Mary's Hospital, Buchon
  - Daejeon St. Mary's Hospital, Daejeon
  - Incheon St. Mary's Hospital, Incheon
  - Seoul St. Mary's Hospital, Seoul
  - St. Mary's Hospital, Seoul
  - Bundang Seoul National hospital, Sungnam
  - Ujeongbu St. Mary's Hospital, Ujeongbu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] De Vita F, Orditura M, Matano E, Bianco R, Carlomagno C, Infusino S, Damiano V, Simeone E, Diadema MR, Lieto E, Castellano P, Pepe S, De Placido S, Galizia G, Di Martino N, Ciardiello F, Catalano G, Bianco AR. A phase II study of biweekly oxaliplatin plus infusional 5-fluorouracil and folinic acid (FOLFOX-4) as first-line treatment of advanced gastric cancer patients. Br J Cancer. 2005 May 9;92(9):1644-9. doi: 10.1038/sj.bjc.6602573. PMID 15856038
- [Background] Park YH, Lee JL, Ryoo BY, Ryu MH, Yang SH, Kim BS, Shin DB, Chang HM, Kim TW, Yuh YJ, Kang YK. Capecitabine in combination with Oxaliplatin (XELOX) as a first-line therapy for advanced gastric cancer. Cancer Chemother Pharmacol. 2008 Apr;61(4):623-9. doi: 10.1007/s00280-007-0515-7. Epub 2007 May 24. PMID 17522863
- [Background] Waddell T, Gollins S, Soe W, Valle J, Allen J, Bentley D, Morris J, Lloyd A, Swindell R, Taylor MB, Saunders MP. Phase II study of short-course capecitabine plus oxaliplatin (XELOX) followed by maintenance capecitabine in advanced colorectal cancer: XelQuali study. Cancer Chemother Pharmacol. 2011 May;67(5):1111-7. doi: 10.1007/s00280-010-1322-0. Epub 2010 Jul 30. PMID 20676676
- [Background] Kang YK, Kang WK, Shin DB, Chen J, Xiong J, Wang J, Lichinitser M, Guan Z, Khasanov R, Zheng L, Philco-Salas M, Suarez T, Santamaria J, Forster G, McCloud PI. Capecitabine/cisplatin versus 5-fluorouracil/cisplatin as first-line therapy in patients with advanced gastric cancer: a randomised phase III noninferiority trial. Ann Oncol. 2009 Apr;20(4):666-73. doi: 10.1093/annonc/mdn717. Epub 2009 Jan 19. PMID 19153121
- [Background] Cunningham D, Starling N, Rao S, Iveson T, Nicolson M, Coxon F, Middleton G, Daniel F, Oates J, Norman AR; Upper Gastrointestinal Clinical Studies Group of the National Cancer Research Institute of the United Kingdom. Capecitabine and oxaliplatin for advanced esophagogastric cancer. N Engl J Med. 2008 Jan 3;358(1):36-46. doi: 10.1056/NEJMoa073149. PMID 18172173
- [Derived] Lee GJ, Kim H, Cho SS, Park HS, An HJ, Woo IS, Byun JH, Hong JH, Ko YH, Sun S, Won HS, Jin JY, Park JC, Kim IH, Roh SY, Shim BY. A Randomized Phase III Study of Patients With Advanced Gastric Adenocarcinoma Without Progression After Six Cycles of XELOX (Capecitabine Plus Oxaliplatin) Followed by Capecitabine Maintenance or Clinical Observation. J Gastric Cancer. 2023 Apr;23(2):315-327. doi: 10.5230/jgc.2023.23.e16. PMID 37129155